CLINICAL TRIAL: NCT03990337
Title: Impact of Ultrasound-guided Identification of Cricoid Cartilage in Cricoid Pressure
Brief Title: Ultrasound-guided Identification of Cricoid Cartilage in Cricoid Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Eric You-Ten, Associate Professor, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 17-0271-A
Record Dates: First submitted 2018-07-30; First posted 2019-06-18 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Endotracheal Intubation; General Anesthesia
Keywords: Ultrasound; Cricoid Cartilage; Cricoid Pressure; General Anesthesia; Endotracheal Intubation
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: prospective two-arm randomized controlled single blinded
Who Masked: Care Provider
Masking Description: Single-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (CPG, n=65) (No Intervention): cricoid pressure applied by the OR nurse on the cricoid cartilage using finger palpation without ultrasonography
- Ultrasound group (USG, n=65) (Active Comparator): cricoid pressure applied by the OR nurse on the cricoid cartilage after localization with ultrasonography
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Ultrasonography of cricoid cartilage.
  Arms: Ultrasound group (USG, n=65)

SUMMARY:
This study is aimed to provide the evidence that ultrasound-guided identification of the cricoid cartilage can improve effectiveness of cricoid pressure. Ultrasound (US) is well recognized as a technique for identifying the neck landmarks including the cricoid cartilage. Based on the potential results that may show that US could be a tool for improve the effectiveness of cricoid pressure, the investigators expect to disseminate this knowledge to be transformed in the standard technique for helping anesthesiologists and nurses to do pressure in the correct location. It is expected that the greatest impact of this study will lead to improved patient outcomes and safety, particularly in the ones with high-risk for aspiration.

DETAILED DESCRIPTION:
This is a prospective two-arm randomized controlled single blinded study to be conducted at Mount Sinai Hospital, University of Toronto. The study will be conducted in the operating rooms (OR) with patients as subjects, and OR nurses and scheduled anesthesiologists as participants.Following signed informed consent, patients will be randomized into two groups:(i) Control group (CPG, n=65): cricoid pressure applied by the OR nurse on the cricoid cartilage using finger palpation without ultrasonography and (ii) Ultrasound group (USG, n=65): cricoid pressure applied by the OR nurse on the cricoid cartilage after localization with US. The oesophagus of the patient participants in both groups will also be identified by US. A portable US machine will be present in the operating room for all patients in both groups.

The anesthesiologist scheduled for the surgery is blinded to group allocation and will induce the patient with general anesthesia. The anesthesiologist will provide adequate oxygenation with 100% oxygen to reach an end-tidal oxygen ≥ 90% using mask ventilation. Thereafter, the scheduled anesthesiologist will step out of the operating room. Apneic oxygenation will be maintained using a nasal cannula with 100% oxygen at 5 litres/min. During apneic oxygenation, one of the research anesthesiologists will localize the cricoid cartilage using US (for patients in USG group). Prior to applying cricoid pressure, the nurse will be instructed to use an estimated pressure (of 30 Newtons) that causes discomfort when applied to his/her nasal bridge. The nurse will then apply an estimated 30 Newtons pressure on the cricoid cartilage localized by US for patients in the USG group or blindly without US for patients in CPG group.

The anesthesiologist will then return to the operating room and perform a videolaryngoscopy to directly visualize up to three attempts to pass a lubricated 20F gastric tube at the upper outlet of the esophagus with (i) pressure directly on the cricoid cartilage and (ii) with pressure on the cricoid cartilage shifted to the left and right of the midline. Following removal of the gastric tube and videolaryngoscope, the trachea will be intubated using direct laryngoscopy with a McIntosh blade. Cricoid pressure will be released after the cuff of the endotracheal tube is inflated. Thereafter, the location of the CC (blindly without US) for patients in CPG group will be marked and compared to the location that will be identified with US.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years,
* ASA physical status I and II,
* body mass index <28 kg/m2,
* scheduled to undergo surgical procedures requiring general anesthesia and endotracheal intubation.

Exclusion Criteria:

* cardiac diseases,
* respiratory diseases,
* liver diseases,
* gastroesophageal reflux symptoms,
* anticipated difficult airway and/or anticipated difficult bag-mask ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2018-07-30 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Cricoid pressure effectiveness | 5 minutes
  Cricoid pressure effectiveness defined as the failure to pass the gastric tube after 3 attempts

SECONDARY OUTCOMES:
Cormack-Lehane classification | 5 minutes
  Cormack-Lehane classification for direct laryngoscopy
Cricoid pressure release | 5 minutes
  necessity of cricoid pressure release for intubation.

CONTACTS AND LOCATIONS:
Overall Officials: Kong Eric You-Ten, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 6 months after publication